CLINICAL TRIAL: NCT02511925
Title: A Pragmatic Crossover Cluster Randomised Study of Electronic Compliance Monitoring of Staff Hand Sanitisation in Critical Care (HANDS Study)
Brief Title: Electronic Hand Hygiene Monitoring and ICU Infection Rates
Acronym: HANDS
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2013IC004B
Record Dates: First submitted 2013-11-26; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Cross Infection
Keywords: Critical care; Feedback
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ICU Cluster 1: Adult Intensive Care Unit - Royal Brompton Hospital
  Interventions: Other: Weekly poster of unit performance; Other: Daily email of personal feedback
- ICU Cluster 2: Paediatric ICU - Royal Brompton Hospital
  Interventions: Other: Weekly poster of unit performance; Other: Daily email of personal feedback; Other: Active reminder from badge
- ICU Cluster 3: Adult Intensive Care Unit - Harefield Hospital
  Interventions: Other: Weekly poster of unit performance; Other: Daily email of personal feedback; Other: Active reminder from badge

INTERVENTIONS:
Other: Weekly poster of unit performance — Weekly feedback is provided to the ICU about current levels of hand hygiene compliance amongst doctors, nurses, and allied healthcare professionals
Other: Daily email of personal feedback — Healthcare workers receive private and personal feedback via email regarding their individual performance benchmarked against the average performance for their professional grouping.
Other: Active reminder from badge — The badge the healthcare worker is wearing vibrates if opportunities to perform hand hygiene are missed
  Groups: ICU Cluster 2; ICU Cluster 3

SUMMARY:
If patients acquire a new infection whilst in hospital this can cause significant morbidity, prolonged hospitalisation and even death. Indeed, there is much public concern about infections such as MRSA. Patients who require intensive care are probably at the greatest risk.

Appropriate hand hygiene by healthcare workers can reduce infection rates and is a key goal of many patient safety initiatives. Worldwide, hand hygiene compliance has been estimated at only 38.7% despite the intervention being simple and cheap. Reasons for poor compliance include lack of time, skin irritation, lack of facilities, intensity of workload and forgetfulness. Furthermore, since cross infection may not be apparent for some days, staff may not associate their (lack of) actions with having caused harm.

Measuring compliance levels enables staff to understand whether they could improve. Direct observation of staff is labour intensive and is not continuous or universal. We will monitor hand hygiene compliance with a newly developed electronic system (MedSense, General Sensing Inc.). We will use the data to provide feedback to the staff in several ways. We hypothesise that comprehensive personalised feedback will reduce healthcare associated infections. We will undertake the study in three intensive care units.

DETAILED DESCRIPTION:
All patients admitted to three intensive care units will be monitored for healthcare associated infections. In parallel the units will be cluster randomised to implement the electronic compliance monitoring in three different ways:

* Unit level feed back every week of current compliance for each of three staff groupings (doctors, nurses, allied health professionals)
* Personalised feedback in the form of an email at the end of a shift stating an individuals performance relative to the average for their professional grouping.
* Real time feedback in the form of a badge worn by the healthcare worker that vibrates when the system thinks they have missed or are about to miss an opportunity for hand hygiene.

All healthcare workers will receive the level of feedback defined in the randomisation for the duration of the three intervention periods. The units will cross-over with an interventing two week wash out period.

All personal feedback will be confidential and private to the individual.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the intensive care units
* All healthcare workers caring for the patients on the intensive care units.

Exclusion Criteria:

* Healthcare workers with skin sensitivity to both alcohol hand rub and soap

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the ICU during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1065 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Composite health care infection rate | Until the end of the second calendar day following ICU discharge
  One of the following three:
  Bacteriological proven infection at a normally sterile site. The sterile sites vein considered are a prior defined as blood, broncho-alveolar lavage, urine sampled from a catheter, chest drain fluid, and surgical wounds. Blood cultures that grow normal skin commensals will be included Endotracheal secretions that culture organisms other than normal upper respiratory tract flora Clostridium difficult related diarrhoea

SECONDARY OUTCOMES:
Incidence of central line associated blood stream infections | Until the end of the second calendar day following ICU discharge
  CDC definition
Incidence of catheter associated urinary tract infections | Until the end of the second calendar day following ICU discharge
  CDC definition
Incidence of ventilator associated pneumonia | Until the end of the second calendar day following ICU discharge
  CDC definition
Incidence of surgical site infection | Until the end of the second calendar day following ICU discharge
  Public Health England definition
Incidence of clostridium difficult diarrhoea | Until the end of the second calendar day following ICU discharge
  Public Health England definition
Incidence of acquisition of new methicilllin resistant staphylococcus aureus | Until the end of the second calendar day following ICU discharge
Incidence of secondary blood stream infections | Until the end of the second calendar day following ICU discharge
  CDC definition
Incidence of antibiotic resistance infections | Until the end of the second calendar day following ICU discharge
  Pre-defined as Acinetobacter baumanii, Pseudomonas aeroginosa (Extended-Spectrum Beta Lacatamase [ESBL] producing), Klebsiella penumoniae (ESBL producing), Escherichia coli (ESBL producing), Stenotrophomonas maltophilia, Serratia marcescens, Clostridium difficile, or MRSA.
Adverse event rate | 24 weeks

OTHER OUTCOMES:
Staff attitudes to electronic compliance monitoring | 0 and 24 weeks
  Quantitative and qualitative analysis of questionnaire data
Surrogate measures of hand hygiene compliance | 24 weeks
  Alcohol hand rub usage, Soap usage and visual compliance monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Cattini, MSc, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Background] Cheng VC, Tai JW, Ho SK, Chan JF, Hung KN, Ho PL, Yuen KY. Introduction of an electronic monitoring system for monitoring compliance with Moments 1 and 4 of the WHO "My 5 Moments for Hand Hygiene" methodology. BMC Infect Dis. 2011 May 26;11:151. doi: 10.1186/1471-2334-11-151. PMID 21612666